CLINICAL TRIAL: NCT03911895
Title: Impact of Stent Length on Short Term Outcomes in Patients With Stable Coronary Artery Disease Undergoing PCI
Brief Title: Impact of Stent Length on Short Term Outcomes in Patients With Stable Coronary Disease Undergoing PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abd elbaset Hassan, Principal investigator, Assiut University
Other Study IDs: Stent length impact on PCI
Record Dates: First submitted 2019-03-26; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Stable Chronic Angina
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- patients with coronary artery diseas undergoing PCI: Effect of stent length on patients with coronary artery undergoing PCI
  Interventions: Device: Stent more than 26 mn length; Device: Stent equal to or less than26 mn length

INTERVENTIONS:
Device: Stent more than 26 mn length — stent length in patients undergoing PCI (Drug Eluting Stent)
Device: Stent equal to or less than26 mn length — stent length in patients undergoing PCI (Drug Eluting Stent)

SUMMARY:
Impact of stent length on short term outcomes in patients with stable coronary artery disease undergoing PCI

DETAILED DESCRIPTION:
Impact of stent length on short term outcomes in patients with stable coronary artery disease undergoing PCI. The investigators will follow up patient clinically and use lab investigation.

ELIGIBILITY:
Inclusion Criteria:

* patient was CAD referred for elective PC as single vessel

Exclusion Criteria:

* patients admitted ACS patients with primary PCI PTCA without stenting No complete revascularization PCI-related coronary complication (diessaction,no really)

Ages: 25 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with stable coronary artery disease undergoing PCI
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Impact of stent length on short term outcomes in patients with stable coronary artery disease undergoing PCI | 3 months
  to study effect of stent length in patients undergoing PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed abdelbast, Asyut, Egypt